CLINICAL TRIAL: NCT05395377
Title: Preventing Diabetes Among Patients With Pre-Diabetes by Improving Patient-Activation and Enhancing Clinical Decision Support for Weight Management to Lower Costs
Brief Title: Preventing Diabetes
Acronym: PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017-0394
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: PreDiabetes
MeSH Terms: conditions — Prediabetic State | interventions — Nutritionists; dentin sialophosphoprotein; Dosage Forms

STUDY DESIGN:
Intervention Model Description: Participants enrolled in this study were able to choose from 1 of 5 intervention options based on their weight status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Registered Dietitian/Nutritionist (Active Comparator)
  Interventions: Behavioral: Registered Dietitian/Nutritionist
- DPP Group Classes (Active Comparator)
  Interventions: Behavioral: Diabetes Prevention Program
- Weight Watchers, Reimagined (Active Comparator)
  Interventions: Behavioral: Weight Watchers, Reimagined
- Pharmacological Treatment (Active Comparator)
  Interventions: Behavioral: DPP or RDN Counseling + Medication
- Bariatric Surgery Evaluation (Active Comparator)
  Interventions: Other: Bariatric Surgery Evaluation

INTERVENTIONS:
Behavioral: Registered Dietitian/Nutritionist — Participants received a FitBit Flex and Intensive Lifestyle Intervention coaching via telephone with Registered Dietitian/Nutritionist.
  Arms: Registered Dietitian/Nutritionist
Behavioral: Diabetes Prevention Program — Modified DPP group classes lead by a Registered Dietitian and Exercise Physiologist.
  Arms: DPP Group Classes
Behavioral: Weight Watchers, Reimagined — Participants in this group were provided with an online access code to enroll in WW and could choose the format of their choice- group, online, and/or smartphone app.
  Arms: Weight Watchers, Reimagined
Behavioral: DPP or RDN Counseling + Medication — Participants met with a weight management specialist to receive weight loss medications, as well as, receiving either the DPP or Registered Dietitian coaching. Medications utilized in this study were Phentermine and Metformin. Metformin was prescribed if the participant could not tolerate Phentermine.
  Arms: Pharmacological Treatment
Other: Bariatric Surgery Evaluation — Participants (BMI > 40) were offered a consultation with the bariatric surgical program that requires lifestyle weight management during the first 6 months. Participants were also able to choose to receive one of the other 4 intervention options in the first six months prior to consideration for bariatric surgery.
  Arms: Bariatric Surgery Evaluation

SUMMARY:
The purpose of this project is to improve the quality of weight management care for patients with pre-diabetes and overweight or obesity. Personalized risk profiles, clinical decision support, and patient-centered decision tools for understanding pre-diabetes risk and the likelihood of preventing diabetes with a modest 5-7% weight loss will be developed. This project will offer patients their choice of effective weight management treatment options, each containing the cornerstone of weight management- intensive lifestyle intervention. Patients and PCPs will be better informed and equipped with information that helps them make weight management treatment decisions that work the best for their lifestyle, and each is expected to produce at least 5-7% weight loss over 6 months.

DETAILED DESCRIPTION:
The primary aim of this study was to demonstrate that an increased recruitment rate for weight loss intervention can be achieved within patients that have pre-diabetes by communicating personalized risk of progression to type 2 diabetes, by estimating risk reduction with weight loss, and by offering program choice. Secondary aims included program participation rate, weight loss, and short term decreased diabetes risk.

ELIGIBILITY:
Inclusion Criteria:

* At least two weight measures within the last two 24 months, including most recent, that meet the following criteria:
* Prediabetes and BMI >27: Treatment Option 1, 2, 3, or 4
* Prediabetes and BMI >40: Treatment Options 1-5
* Most recent laboratory value that meets prediabetes indicators, per American Diabetes Association, 2016
* Hemoglobin A1C ≥5.7% and <6.5%, or
* Fasting plasma glucose ≥100 mg/dl and <126 mg/dl, or
* Oral glucose tolerance test ≥140 mg/dl and <200 mg/dl

Exclusion Criteria:

* History of significant weight loss documented within 5 years,
* Contraindications to weight change (e.g., cancer, pregnancy)
* Prior bariatric surgery
* Weight loss medication use or orders within 5 years prior to the project.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2021-11-16 (Actual)

PRIMARY OUTCOMES:
Demographics | Baseline
  Race, ethnicity, education level, marital status, household income, and weight management history.
Body Weight | 12 Months
  The study's primary outcome is change in body mass index (in kg) from baseline to 12-month follow-up.
Pre-Diabetes Indicator | 12 months
  At baseline, 6 months,12 months, we will assess HbA1c from the intervention participants. These measures will provide important information about changes in participants' risk and prevention of diabetes.
Patient-Centered Outcomes | 12 months
  Treatment satisfaction and patient involvement in care survey

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Bailey-Davis, DEd, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Health System, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No